CLINICAL TRIAL: NCT00907933
Title: A Randomized, Double-blind, Placebo-controlled Study in Healthy Volunteers to Examine the Safety, Tolerability and Pharmacokinetics of a) Single, Ascending and b) Twice-daily Repeat Doses of Intranasal SB-705498
Brief Title: Intranasal SB-705498 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 111610
Record Dates: First submitted 2009-04-30; First posted 2009-05-25 (Estimated); Last update posted 2017-07-13 (Actual); Status verified 2017-07

CONDITIONS: Rhinitis
MeSH Terms: conditions — Rhinitis | interventions — SB 705498

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (9):
- Part 1 - Arm 1 (Experimental): HVTs
  Interventions: Drug: SB-705498
- Part 2 - Arm 3 (Placebo Comparator): HVTs
  Interventions: Drug: Placebo
- Part 1 - Arm 2 (Experimental): HVTs
  Interventions: Drug: SB-705498
- Part 1 - Arm 3 (Experimental): HVTs
  Interventions: Drug: SB-705498
- Part 1 - Arm 4 (Experimental): HVTs
  Interventions: Drug: SB-705498
- Part 1 - Arm 5 (Experimental): HVTs
  Interventions: Drug: SB-705498
- Part 1 - Arm 6 (Placebo Comparator): HVTs
  Interventions: Drug: Placebo
- Part 2 - Arm 1 (Experimental): HVTs
  Interventions: Drug: SB-705498
- Part 2 - Arm 2 (Experimental): HVTs
  Interventions: Drug: SB-705498

INTERVENTIONS:
Drug: SB-705498 — 0.5mg intranasal SB-705498
  Arms: Part 1 - Arm 1
Drug: SB-705498 — 1.5mg intranasal SB-705498
  Arms: Part 1 - Arm 2
Drug: SB-705498 — 3mg intranasal SB-705498
  Arms: Part 1 - Arm 3
Drug: SB-705498 — 6mg intranasal SB-705498
  Arms: Part 1 - Arm 4
Drug: SB-705498 — 12mg intranasal SB-705498
  Arms: Part 1 - Arm 5
Drug: Placebo — Placebo '498
  Arms: Part 1 - Arm 6
Drug: SB-705498 — 6mg intranasal SB-705498 for 14 days bid
  Arms: Part 2 - Arm 1
Drug: SB-705498 — 12mg intranasal SB-705498 14 days bid
  Arms: Part 2 - Arm 2
Drug: Placebo — Placebo
  Arms: Part 2 - Arm 3

SUMMARY:
This is a First Time in Human (FTIH) study to investigate the safety, tolerability and pharmacokinetics (PK) of a) single, escalating and b) twice-daily 14 days repeat doses of intranasal SB-705498 in healthy volunteers (HVT). The safety and tolerability of single intranasal 498 dosing will be assessed and established before initiating the evaluation of repeat intranasal 498 dosing.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, as determined by a responsible physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring.
* Male or female between 18 and 60 years of age inclusive.
* A female subject is eligible to participate if she is of:
* Non-childbearing potential defined as females with documented tubal occlusion, bilateral salpingectomy, bilateral oophorectomy or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous FSH > 40 MlU/ml and estradiol < 40 pg/ml (<140 pmol/L) is confirmatory]. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the contraception methods in the protocol if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrolment. For most forms of HRT, at least 2-4 weeks should elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT. Following confirmation of their post-menopausal status, they can resume use of HRT during the study without use of a contraceptive method.
* Child-bearing potential and agrees to use one of the contraception methods listed in the protocol. Female subjects willing to participate in the study must agree to use contraception from the screening visit until 15 days post-last treatment administration.
* Male subjects must agree to use one of the contraception methods listed in the protocol. For male subjects willing to participate in the study this criterion must be followed from the time of the screening visit until 15 days post-last treatment administration.
* Non-smoker for at least 6 months with a pack history less than or equal to 5 pack years (Pack years = (No. of cigarettes smoked/day/20) x No. of years smoked).
* Body weight greater than or equal to 50 kg and body mass index (BMI) within the range 19 - 29.9 kg/m2 (inclusive).
* Normal assessment of vital signs and 12-lead ECG at screening. A subject may be included in the study if any abnormality is deemed not clinically significant by the Investigator.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* Available to complete all the required study measurements.

Exclusion Criteria:

* Past medical history of rhinitis, including allergic, non-allergic rhinitis and rhinosinusitis. Subjects with recent upper respiratory tract infections (URTIs) will be allowed in the study only if their nasal symptoms have been completely resolved for more than 3 weeks prior to screening.
* Nasal conditions likely to affect the outcome of the study, i.e. nasal septal perforation, nasal polyps, other nasal malformations.
* History of frequent nosebleeds.
* A history of gastro-intestinal, hepatic, renal or other condition known to interfere with the absorption, distribution, metabolism or excretion of drugs.
* History of regular alcohol consumption within 6 months of the study defined as: an average weekly intake of greater than 21 units or an average daily intake of greater than 3 units (males), or defined as an average weekly intake of greater than 14 units or an average daily intake of greater than 2 units (females). One unit is equivalent to a half-pint (220mL) of beer or 1 (25ml) measure of spirits or 1 glass (125ml) of wine.
* Positive pre-study drug/alcohol/smoking screen. A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine, opiates, cannabinoids, benzodiazepines and methadone.
* Positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* A positive test for human immunodeficiency virus (HIV) antibody.
* Exposure to more than four new chemical entities within 6 months prior to the start of the study.
* Participation in a clinical trial with a new molecule entity or any other clinical trial within 3 months of the start of the study.
* Use of prescription or non-prescription drugs, as well as of vitamins, herbal and dietary supplements (including St John's Wort) within 7 days prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* History of drug or other allergy that, in the opinion of the Investigator or GSK Medical Monitor, contraindicates participation in this study.
* Donation of blood or blood products in excess of 500mL within a 56 day period prior the start of this study.
* Pregnant females as determined by positive serum or urine beta-human chorionic gonadatrophin (beta-hCG) test at screening or prior to dosing.
* Lactating females.
* Unwillingness or inability to follow the procedures outlined in the protocol.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2008-11-10 (Actual); Primary Completion 2009-02-11 (Actual); Study Completion 2009-02-11 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability (Electrocardiogram, vital signs, lab tests, AEs and nasal tolerability | Various

SECONDARY OUTCOMES:
Part 1: Single dose derived pharmacokinetics (Cmax, tmax, AUC(0-4) and AUC(o-infinity); Part 2: Repeat dose derived pharmacokinetics (Cmax, tmax, AUC(0-4) and AUC(o-infinity) | Part 1: Various timepoints through the day; Part 2: Various timepoints over 14 days

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study 111610 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/111610?search=study&search_terms=111610#rs
- Available data/document: Study Protocol: 111610 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 111610 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 111610 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 111610 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 111610 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 111610 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 111610 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register